CLINICAL TRIAL: NCT04862793
Title: Impact of Computerized Feedback During Colonoscopy on Adenoma Detection Rate of Colorectal Cancer and Patient Related Satisfaction: A Cluster-randomized Controlled Trial.
Brief Title: Computerized Feedback in Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Collaborators: Danish Cancer Society (Other); Ambu A/S (Industry); Region Capital Denmark (Other); Herlev Hospital (Other); Bispebjerg Hospital (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Kristoffer Mazanti Cold, Principal Investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P-2021-256
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Healthy
Keywords: Colonoscopy; Adenoma Detection Rate; Computerized Feedback
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized controlled cluster trial following a stepped-wedge randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback (Experimental): Feedback system through CoPS and CoRS
  Interventions: Device: Colonoscopy Progression Score (CoPS); Device: Colonoscopy Retraction Score (CoRS)
- Standard procedure (No Intervention): Performing the standard procedure in accordance with the departments usual conduct.

INTERVENTIONS:
Device: Colonoscopy Progression Score (CoPS) — The Colonoscopy Progression Score consists of five different aspects: Travel length, Tip progression, chase efficiency, shaft movement without tip progression and looping.
  Arms: Feedback
Device: Colonoscopy Retraction Score (CoRS) — The Colonoscopy Retraction Score consists of three different aspects: Tip Retraction, Retraction Efficiency, and Retraction Distance.
  Arms: Feedback

SUMMARY:
In a cluster-randomized study compare if feedback from two computerized feedback systems doing a colonoscopy (CoPS and CoRS) can improve the adenoma detection rate and decrease patient discomfort.

DETAILED DESCRIPTION:
Background:

Approximately 4,600 persons get colon cancer annually in Denmark and it is the second most common cause of cancer death. Survival is highly dependent on early detection through a colonoscopy. A thorough colonoscopy is essential to detect early cancers but unfortunately the quality of colonoscopies varies widely between operators. A study of 314,872 colonoscopies performed by 136 gastroenterologists found that the adenoma detection rate (ADR) ranged from 7 - 53% and was inversely associated with the risks of fatal interval cancer. The investigators have developed to tools that can generate automatic, computerized feedback in order to make a more thorough procedure and reduce patient discomfort, the Colonoscopy Progression Score (CoPS) and Colonoscopy Retraction Score (CoRS)

Objectives:

The investigators predict that live-feedback from CoPS and CoRS doing a colonoscopy can improve the ADR and subsequent prevent colorectal cancer. The aim of this project is to:

1. In a cluster-randomized study compare if feedback from CoPS and CoRS can improve the adenoma detection rate and patient satisfaction for individual operators and the department as a whole.
2. Make an immediate measure to assess the quality of individual colonoscopy performance.

Materials and methodology:

As a randomized controlled cluster trial following a stepped-wedge program, feedback doing a colonoscopy from these (CoPS and CoRS) will be tested compared to no feedback. Three test departments consisting of three University Hospital in the Capital region of Denmark will be included.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for a screening colonoscopy through the Danish National Screening Program for Colorectal Cancer.

Exclusion Criteria: Incomplete procedure due to:

* In cases were the cecum is not reached.
* Unsatisfactory bowel preparation which results in admission for a new procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feedback from CoRS results in change in Adenoma Detection Rate for individual operators and for the department as a whole. | Baseline (pre-intervention) and with the end of each time cluster (month 8, 12, 16, 18). The intervention will be at different time clusters for the three participating hospitals, and therefore the baseline sampling period will be different.
  The Adenoma Detection Rate of an operator is correlated to patient survival of colorectal cancer. A low Adenoma Detection Rate is correlated with a higher occurrence of interval cancer. Increasing the Adenoma Detection Rate will result in a more beneficial screening program with more cancers being caught in an earlier state and thereby increase patient survival.
Feedback from CoPS results in change in patient discomfort. | Baseline (pre-intervention) and with the end of each time cluster (month 8, 12, 16, 18). The intervention will be at different time clusters for the three participating hospitals, and therefore the baseline sampling period will be different.
  Patient discomfort will be assessed by a post-procedure questionnaire. We will examine the correlation between the intervention and patient discomfort, and assess if more procedures can be completed due to less patient discomfort using the intervention.

SECONDARY OUTCOMES:
Make an immediate measure to assess the quality of individual colonoscopy performance. | On data collection completion, estimated December 2023
  To measure a reliable Adenoma detection rate, 500 procedures are needed. We will aim to make an immediate measure based on CoRS to assess the quality of each colonoscopy and investigate this measures correlation to the ADR in the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Mazanti Cold, MD, Principal Investigator — PhD-alumni

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At end of data collection (December 2023) and for the following 5 years.
Access Criteria: On request to the primary investigator with a useful scientific purpose.